CLINICAL TRIAL: NCT00679159
Title: A Phase II Study Evaluating the Safety and Immunogenicity of a New TB Vaccine, MVA85A, in Healthy Children and Infants After BCG Vaccination at Birth
Brief Title: A Study of MVA85A in Healthy Children and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB014; MCC: 20070156
Record Dates: First submitted 2008-04-02; First posted 2008-05-16 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A; MVA Pfs25-IMX313 malaria vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): 24 children (5 x 10^7pfu)
  Interventions: Biological: MVA85A
- 2 (Experimental): 36 infants (2.5 x 10^7pfu)
  Interventions: Biological: MVA85A
- 3 (Experimental): 36 infants (5 x 10^7 pfu)
  Interventions: Biological: MVA85A
- 4 (Experimental): 36 infants (1 x 10^8pfu)
  Interventions: Biological: MVA85A
- 5 (Placebo Comparator): 36 infants (Prevenar vaccine)
  Interventions: Biological: Prevenar

INTERVENTIONS:
Biological: MVA85A — Modified vaccinia virus Ankara expressing antigen 85A from M. tuberculosis
  Other Names: Modified vaccinia virus Ankara
  Arms: 1; 2; 3; 4
Biological: Prevenar — Streptococcus pneumoniae vaccine
  Arms: 5

SUMMARY:
This study is designed to evaluate the safety of the TB vaccine MVA85A in healthy children and infants in South Africa. A single vaccination with MVA85A has been shown to be safe and highly immunogenic in a wide range of subjects in previous clinical trials. In this trial,we will vaccinate 24 children with 5 x 10^7pfu of MVA85A and three groups of 36 infants with 2.5 x 10^7, 5 x 10^7 or 1 x 10^8 pfu.

Participants will be identified from the general population living in Worcester, Western Cape, South Africa

DETAILED DESCRIPTION:
M.tb is an intracellular organism and protective immunity is dependent on an intact cellular immune system. Both Class II-restricted CD4+ and Class I-restricted CD8+ T lymphocytes are important for protection. Gamma delta cells and non-classically restricted T cells such as CD1-restricted T cells may also play a protective role but knowledge of how to induce these to protective levels by vaccination is very limited. Although several vaccine delivery systems are capable of inducing T cells, e.g. protein/adjuvant combinations, DNA vaccines and recombinant viral vectors, when used alone these delivery systems induce only low-level responses. Heterologous prime-boost immunisation strategies involve immunizing with 2 two different vaccines, each expressing the same antigen, several weeks apart. These strategies induce higher levels of CD4+ and CD8+ T cells than homologous boosting in animal models of malaria, HIV and TB.

Recombinant modified vaccinia virus Ankara expressing antigen 85A (MVA85A). When used in heterologous prime-boost strategies, some viral vectors are very good at boosting previously primed T cell responses, particularly recombinant adenoviral constructs and recombinant pox viruses. Modified vaccinia virus Ankara (MVA) is an attenuated strain of vaccinia virus that has been passaged more than 500 times through chick embryo fibroblasts and as a consequence has lost both host range genes and cytokine receptor genes. MVA has an excellent safety record, as it was used to vaccinate more than 120,000 people at the end of the smallpox eradication campaign, with no serious adverse events. In humans, several hundred HIV negative volunteers have now been immunized with recombinant MVAs expressing a number of different antigens, with no serious adverse events. A recombinant MVA expressing an antigen from Plasmodium falciparum has been demonstrated to boost CD4+ and CD8+ T cells in humans. Recombinant MVAs are now in clinical trials for several infectious diseases including HIV, hepatitis B and malaria. Importantly, for a new TB vaccine, the safety of MVA as a viral vector has now been demonstrated in HIV positive patients.

Including BCG in such heterologous prime-boost regimes allows for the beneficial effects of BCG to be retained. We have developed an immunisation strategy using BCG as the priming immunisation and a recombinant MVA (rMVA) as the boost. The antigen selected for inclusion in the rMVA must be present in all strains of BCG. We have selected Antigen 85A, which forms part of the immunodominant antigen 85 complex. Although there are numerous candidate antigens for use in a TB vaccine, antigen 85A has long been considered a leading choice. It is a major target antigen recognised by T cells from infected individuals and it is protective as a DNA vaccine in small animals. Importantly, for use in BCG prime-MVA boost regimes, it is highly conserved amongst all mycobacterial species and is present in all strains of BCG. In small animals it is a major target of the immune responses induced by BCG and in humans HLA-A2 restricted CD8 T cells have been found in a high proportion of BCG-immunised individuals. Antigen 85A is an enzyme, mycolyl transferase, which is involved in cell wall biosynthesis.

Pre-clinical data Using this BCG prime-MVA85A boost in BALB/c mice induces higher levels of both antigen specific interferon-gamma (IFN-γ) secreting CD4 T and CD8+ T cells and higher levels of protection than after BCG alone. This regime has now been further evaluated in the more sensitive guinea pig aerosol challenge model with very encouraging results. Guinea pigs vaccinated with BCG, followed by MVA85A, and then further boosted with a second recombinant viral vector, fowlpox, expressing antigen 85A (FP85A) showed significantly greater protection against challenge than guinea pigs vaccinated with BCG alone. This regime is also immunogenic and protective in rhesus macaques

Clinical studies The safety and immunogenicity of this BCG prime-MVA85A boost vaccination strategy has now been evaluated in a series of small-scale Phase I studies in the UK. MVA85A was the first candidate TB vaccine in clinical trials anywhere in the world in September 2002, and is currently the only one in clinical trials in Africa . The main immunological read-out used in these clinical trials is the ex-vivo IFN-γ Elispot assay, which is used to assess specific T cell responses to tuberculin PPD, antigen 85 complex and pools of overlapping peptides spanning the length of antigen 85A. The best immunological correlate of protection in murine and human TB is the secretion of IFN-γ from sensitised T cells.

In the UK, 14 mycobacterially and BCG naïve, healthy volunteers have been vaccinated with 5 x 10^7pfu MVA85A, administered intradermally. We find that MVA85A is safe and well tolerated. A single vaccination with MVA85A induces remarkably high levels of specific effector T cell responses (median IFN- γ Elispot response to Antigen 85A summed peptide pools 1153 spots per million PBMC). In addition, the safety of MVA85A in volunteers previously vaccinated with BCG has now been demonstrated in 17 volunteers. These 17 volunteers show even higher peak levels of antigen specific T cells (median response 2455 spots per million PBMC) 1 week post-vaccination than those immunized with MVA85A alone. Perhaps more importantly for the induction of T cell memory, volunteers who have been previously BCG vaccinated maintain higher levels of antigen specific T cells after MVA85A for up to 24 weeks after vaccination, when compared to those volunteers vaccinated with MVA85A alone. In contrast to this viral vector boost, the magnitude of T cell responses seen after vaccination with a leading protein/adjuvant vaccine (for malaria), RTS,S/AS02, is around 200 spots per million PBMC.

This series of Phase I studies have also replicated in The Gambia, and the results from The Gambia are equally promising. In both the UK and The Gambian studies, MVA85A induces 5-10 fold higher immune responses than any other recombinant MVA in clinical trials. The most likely explanation for this is that the volunteers have some weak pre-existing anti-mycobacterial immunity induced by exposure to environmental mycobacteria, and this specific anti-mycobacterial immunity is being boosted by MVA85A. We have some preliminary data to support this hypothesis, and other groups have also found pre-existing immunity to environmental mycobacteria in healthy UK adults. Vaccines that are good at boosting previously primed T cell responses, such as MVA85A, are potentially good candidates for a post-exposure vaccine designed to boost the immune response and prevent the development of disease in those latently infected. If the high levels of specific T cells seen after a single immunisation with MVA85A are attributable to the boosting of pre-existing environmentally induced responses, then this makes MVA85A an extremely promising candidate for a boosting vaccine, given as a post-exposure vaccine in latent infection.

The next study, which completed enrolment in the UK in February 2006, assessed the safety and immunogenicity of MVA85A in healthy volunteers who were latently infected with M.tb. Twelve latently infected healthy subjects were vaccinated with a single dose of 5 x 10^7pfu MVA85A. In this study, latent M.tb infection was determined by tuberculin skin testing and ex-vivo IFN-γ Elispot responses to two M.tb specific antigens, ESAT6 and CFP10. Follow-up involved detailed radiological and clinical assessment of the safety of this vaccine in M.tb infected subjects. We found that MVA85A is equally safe and equally immunogenic in this latently infected population as it is in the population vaccinated with BCG (Sander et al, unpublished data). We have also conducted a dose finding study looking at two further doses of MVA85A, 1 x 10^7pfu and 1 x 10^8 pfu. Twelve subjects were vaccinated with each dose. The preliminary results show the vaccine is significantly more immunogenic at the higher (1 x 10^8 pfu) dose but the immunogenicity of the lower (1 x 10^7 pfu) dose is comparable with the standard (5 x 10^7pfu) dose.

We have just started enrolment into an HIV study where antiretroviral naïve, HIV infected adults with a CD4 count greater than 350 are vaccinated with MVA85A. To date, there have been no safety concerns with this study.

MVA85A is being trialled in a series of Phase I and II studies in the Western Cape province, South Africa, where the prevalence of tuberculosis is extremely high (annual incidence of disease ~1%). In August 2005, enrolment commenced into trial 008 and it continued until July 2006. 24 healthy TB naïve and HIV uninfected adults were vaccinated. The preliminary results of this arm of the trial were presented in Vienna (Hawkridge et al, TB Vaccines for the World; April 2006) and Paris the vaccine was shown to be safe and highly immunogenic. Enrolment into the adolescent arm of this study commenced in November 2006 once it was clear that the day 84 safety results in the adults were satisfactory.

This protocol forms the second part of these age de-escalation studies in South Africa, which are necessary before we commence a Phase IIb proof-of-concept efficacy trial with MVA85A in this population in 2008.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be children or infants aged 6 months - 11 years.
* Subject's parent/guardian is willing and able to give written informed consent for participation in the study.
* Subject is BCG vaccinated within the first 4 weeks of life
* In addition, informed assent will be obtained from all children aged 7 years or older unless they are adjudged incapable of understanding the basic concepts covered in the informed assent form, and an attempt will be made to obtain informed assent from children aged younger than 7 years if they are judged capable of understanding the basic concepts covered in the informed assent form
* Subject is in good health
* Subject has clinically acceptable laboratory results from screening visit
* CXR normal with no evidence of active or past TB
* Subject's parent/legal guardian is willing to allow child to undergo an HIV test
* Parent/guardian and subject able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Subject is Mantoux (>10 mm) and/or ELISPOT (> 50 spots/million PBMC) positive for M tb (PPD, ESAT 6 and/or CFP10)
* Subject is HIV antibody positive
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patient/subject at risk because of participation in the study, or may influence the result of the study, or the patient/subject's ability to participate in the study.
* Patient/subjects/healthy volunteers who have participated in another research study involving an investigational product in the past 12 weeks
* Patient/subjects previously enrolled into this study.
* Received a live vaccine (e.g. measles) in the previous 4 weeks or due to receive a live vaccine in the 4 weeks following enrolment

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety of MVA85A. Both local and systemic adverse events will be monitored, including a daily diary card for the first week. Blood will be taken at day 7 and day 28 for biochemistry and haematology. | 3 months

SECONDARY OUTCOMES:
Immunogenicity of MVA85A | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford; Gregory Hussey, Principal Investigator — University of Cape Town
Locations (1):
- University Cape Town, Worcester, Western Cape, South Africa

REFERENCES:
- [Derived] Scriba TJ, Tameris M, Mansoor N, Smit E, van der Merwe L, Mauff K, Hughes EJ, Moyo S, Brittain N, Lawrie A, Mulenga H, de Kock M, Gelderbloem S, Veldsman A, Hatherill M, Geldenhuys H, Hill AV, Hussey GD, Mahomed H, Hanekom WA, McShane H. Dose-finding study of the novel tuberculosis vaccine, MVA85A, in healthy BCG-vaccinated infants. J Infect Dis. 2011 Jun 15;203(12):1832-43. doi: 10.1093/infdis/jir195. PMID 21606542